CLINICAL TRIAL: NCT00098345
Title: An Open Label, Two Stage, Phase II Study to Evaluate the Efficacy and Tolerability of ZD6474 in Patients With Locally Advanced or Metastatic Hereditary Medullary Thyroid Carcinoma.
Brief Title: Efficacy and Tolerability of ZD6474 in Patients With Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00008; LPS14954 (Other: Sanofi)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Results first posted 2011-05-24 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Thyroid Cancer
Keywords: Caprelsa (vandetanib); ZD6474
MeSH Terms: conditions — Thyroid Neoplasms | interventions — vandetanib

ARMS (1):
- Caprelsa (vandetanib) 300 mg (Experimental): Daily oral dose of Caprelsa (vandetanib) 300mg
  Interventions: Drug: ZD6474 (vandetanib)

INTERVENTIONS:
Drug: ZD6474 (vandetanib) — oral once daily tablet
  Other Names: Caprelsa™ (vandetanib); SAR390530

SUMMARY:
The purpose of this open label, two stage, phase II study is to evaluate the efficacy and tolerability of ZD6474 in patients with locally advanced or metastatic hereditary medullary thyroid carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or hereditary medullary thyroid cancer
* Signed informed consent
* One or more measurable lesions

Exclusion Criteria:

* Brain metastases or spinal cord compression
* Specific laboratory ranges
* Specific heart problems
* Prior chemotherapy and/or radiation therapy
* Participation in other trials within 30 days

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-11; Primary Completion 2008-02 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (5):
  - Research Site, San Francisco, California
  - Research Site, New Haven, Connecticut
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Houston, Texas
- Research Site, Villejuif, France

REFERENCES:
- [Background] Wells SA Jr, Gosnell JE, Gagel RF, Moley J, Pfister D, Sosa JA, Skinner M, Krebs A, Vasselli J, Schlumberger M. Vandetanib for the treatment of patients with locally advanced or metastatic hereditary medullary thyroid cancer. J Clin Oncol. 2010 Feb 10;28(5):767-72. doi: 10.1200/JCO.2009.23.6604. Epub 2010 Jan 11. PMID 20065189
- See also: CSR-D4200C00008.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=339&filename=CSR-D4200C00008.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 12 November 2004, last patient enrolled 15 August 2006, cut off date 22 February 2008. 40 patients were enrolled in the study.
Pre-assignment Details: 40 patients were enrolled/screened to the study but only 30 patients were entered treatment/randomized.
Period: Overall Study
Arm/Group | Caprelsa (Vandetanib) 300 mg
Started | 30
Completed | 17 (ongoing study treatment at data cut-off)
Not Completed | 13
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 2
Not completed — progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | Caprelsa (Vandetanib) 300 mg
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 48.7 [20 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The ORR is the number of patients that are responders ie those patients with a confirmed best objective response of complete response (CR) or partial response (PR) defined according to RECIST 1.0.
Time Frame: Pre-dose and every 12 weeks up to RECIST progression as defined according to RECIST 1.0.
Measure: Number; unit: Participants
Arm/Group | Caprelsa (Vandetanib) 300 mg
Number analyzed (Participants) | 30
Participants | 6

2. Secondary Outcome: Progression Free Survival
Description: Median time to progression defined according to RECIST 1.0 (months) from randomisation until objective disease progression or death (by any cause in the absence of objective progression) provided death is within 3 months from the last evaluable RECIST assessment.
Time Frame: Pre-dose and every 12 weeks up to RECIST progression as defined according to RECIST 1.0.
Population: Upper limit is a censored value
Measure: Median (Full Range); unit: months
Arm/Group | Caprelsa (Vandetanib) 300 mg
Number analyzed (Participants) | 30
months | 27.9 [2.56 to 36.11]

3. Secondary Outcome: Duration of Objective Response
Description: Median duration of objective response as defined according to RECIST 1.0 from onset of response until data of objective disease progression or death from any cause in days.
Time Frame: Pre-dose and every 12 weeks up to RECIST progression as defined according to RECIST 1.0.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Caprelsa (Vandetanib) 300 mg
Number analyzed (Participants) | 30
days | 310.5 [245 to 402]

4. Secondary Outcome: Disease Control Rate
Description: Disease control rate was defined as the number of patients who had a best response of Complete Response (CR), or Partial Response (PR) or stable disease (SD) ≥24 weeks as defined according to RECIST 1.0.
Time Frame: Pre-dose and every 12 weeks up to RECIST progression as defined according to RECIST 1.0.
Measure: Number; unit: Participants
Arm/Group | Caprelsa (Vandetanib) 300 mg
Number analyzed (Participants) | 30
Participants | 22

5. Secondary Outcome: Biochemical Response Calcitonin (CTN)
Description: A patient's best biochemical response was calculated from assessments performed at baseline and during treatment. Responders were those patients with a confirmed best biochemical response of Complete Response or Partial (i.e. complete normalization of CTN or at least a 50% decrease in CTN from baseline).
Time Frame: Blood samples for analysis of CTN taken on Day 1 (every 3 hours for 24 hours), then a single sample on Day 5, weekly through the first 2 assessment periods, monthly (prior to amendment 7) and every 12 weeks (following amendments) until discontinuation
Measure: Number; unit: Participants
Arm/Group | Caprelsa (Vandetanib) 300 mg
Number analyzed (Participants) | 30
Participants | 24

6. Secondary Outcome: Symptomatic Response
Description: Number of participants with a reduction of frequency and improvement in consistency of stool to normal (no more than 2 solid stools daily without concomitant anti-diarrheal medication) following administration of Caprelsa (vandetanib) denoted a symptomatic CR. An improvement in stool consistency to mostly semisolid and decrease in stool frequency to 50% or greater denoted symptomatic PR.
Time Frame: Symptomatic diarrhea was assessed using stool frequency and consistency diaries. Baseline was established using the average of the 4 days immediately prior to first dose on Day 5. Diaries were completed every day for the first 6 months on study drug.
Measure: Number; unit: Participants
Arm/Group | Caprelsa (Vandetanib) 300 mg
Number analyzed (Participants) | 30
Participants | 0

7. Secondary Outcome: World Health Organisation (WHO) Performance Status
Description: Number of patients demonstrating a worsening (increase in score of one or more from baseline) in WHO PS from baseline to 24 weeks. WHO PS is scored zero (Fully active) to 4 (completely disabled)
Time Frame: Performance status was assessed using the WHO criteria at baseline and because SD lasting for at least 24 weeks was used in the definition of disease control (in addition to confirmed objective response), WHO PS at 24 weeks was evaluated.
Measure: Number; unit: Participants
Arm/Group | Caprelsa (Vandetanib) 300 mg
Number analyzed (Participants) | 30
Participants | 4

ADVERSE EVENTS:
Description: Other (non-serious) adverse events terms were reported as per MedDRA 11.0.
Arm/Group | Caprelsa (Vandetanib) 300 mg
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 14/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caprelsa (Vandetanib) 300 mg (N=30)
Cardiac Failure (Cardiac disorders) | 1
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pancreatitis Acute (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Abdominal Infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Diverticulitis Intestinal Haemorrhagic (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Electrocardiogram Qt Prolonged (Investigations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Hot Flush (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Caprelsa (Vandetanib) 300 mg (N=30)
Anaemia (Blood and lymphatic system disorders) | 3
Bradycardia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 2
Conjunctivitis (Eye disorders) | 2
Dry Eye (Eye disorders) | 2
Vision Blurred (Eye disorders) | 7
Visual Disturbance (Eye disorders) | 3
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 21
Dry Mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 19
Oesophagitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 6
Chest Discomfort (General disorders) | 2
Chills (General disorders) | 5
Face Oedema (General disorders) | 2
Fatigue (General disorders) | 19
Influenza Like Illness (General disorders) | 2
Localised Oedema (General disorders) | 2
Mucosal Inflammation (General disorders) | 3
Oedema (General disorders) | 2
Oedema Peripheral (General disorders) | 7
Pyrexia (General disorders) | 4
Temperature Intolerance (General disorders) | 6
Bronchitis (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 2
Paronychia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Upper Respiratory Tract Infection (Infections and infestations) | 4
Urinary Tract Infection (Infections and infestations) | 7
Contrast Media Reaction (Injury, poisoning and procedural complications) | 2
Blood Alkaline Phosphatase Increased (Investigations) | 2
Blood Creatinine Increased (Investigations) | 3
Blood Urea Increased (Investigations) | 2
Electrocardiogram Qt Prolonged (Investigations) | 7
Platelet Count Increased (Investigations) | 2
Weight Decreased (Investigations) | 4
Weight Increased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 13
Decreased Appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 10
Dyskinesia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 14
Paraesthesia (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 6
Haematuria (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 2
Urinary Retention (Renal and urinary disorders) | 3
Menstruation Irregular (Reproductive system and breast disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 6
Acne (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 4
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 9
Erythema (Skin and subcutaneous tissue disorders) | 2
Periorbital Oedema (Skin and subcutaneous tissue disorders) | 2
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 20
Rash Erythematous (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 3
Hot Flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.